CLINICAL TRIAL: NCT02368886
Title: Regorafenib Dose Optimization Study (ReDOS): A Phase II Randomized Study of Lower Dose Regorafenib Compared to Standard Dose Regorafenib in Patients With Refractory Metastatic Colorectal Cancer (mCRC)
Brief Title: Lower or Standard Dose Regorafenib in Treating Patients With Refractory Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RU021407I; NCI-2015-00011 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU021407I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Colon Adenocarcinoma; Rectal Adenocarcinoma; Stage III Colorectal Cancer AJCC v7; Stage IIIA Colorectal Cancer AJCC v7; Stage IIIB Colorectal Cancer AJCC v7; Stage IIIC Colorectal Cancer AJCC v7; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Clobetasol; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A1 (lower-dose regorafenib, pre-emptive clobetasol) (Experimental): Patients receive lower-dose regorafenib PO QD on days 1-21 and pre-emptive clobetasol propionate given topically BID for 12 weeks, beginning on day 1 of regorafenib.
  Interventions: Drug: Clobetasol Propionate; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Drug: Regorafenib
- Arm A2 (lower-dose regorafenib, reactive clobetasol) (Experimental): Patients receive lower-dose regorafenib PO as in Arm A1 and reactive clobetasol propionate given topically BID beginning on day 1 per physician discretion upon occurrence of PPES grade >= 1.
  Interventions: Drug: Clobetasol Propionate; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Drug: Regorafenib
- Arm B1 (standard dose regorafenib, pre-emptive clobetasol) (Experimental): Patients receive standard dose regorafenib PO QD on days 1-21 and pre-emptive clobetasol propionate as in Arm A1.
  Interventions: Drug: Clobetasol Propionate; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Drug: Regorafenib
- Arm B2 (standard dose regorafenib, reactive clobetasol) (Experimental): Patients receive standard dose regorafenib PO as in Arm B1 and reactive clobetasol propionate as in Arm A2.
  Interventions: Drug: Clobetasol Propionate; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Drug: Regorafenib

INTERVENTIONS:
Drug: Clobetasol Propionate — Given topically
  Other Names: Olux-E
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Stivarga

SUMMARY:
This randomized phase II trial studies how well lower-dose compared to standard dose regorafenib works in treating patients with colorectal cancer that has spread from the primary site (place where it started) to other places in the body and does not respond to treatment. Regorafenib may stop the growth of colorectal cancer by blocking the growth of new blood vessels necessary for tumor growth and by blocking some of the enzymes needed for cell growth. It is not yet known whether lower-dose or standard dose regorafenib is more effective in treating patients with colorectal cancer. Clobetasol propionate is a steroid cream that is commonly used to treat a variety of skin conditions and may help prevent hand-foot skin reactions in patients receiving regorafenib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the proportion of patients who complete 2 cycles of protocol treatment and initiate cycle 3 in arm A (pooled arm A1 and A2) and arm B (pooled arm B1 and B2).

SECONDARY OBJECTIVES:

I. Evaluate outcome measures for efficacy in each arm including progression-free survival (PFS), time to progression (TTP), and overall survival (OS).

II. Compare between arms the cumulative dose and dose intensity received within the first two cycles.

III. Evaluate the proportion of patients in each arm that exhibit grade 3 palmar-plantar erythrodysesthesia syndrome (PPES) and/or fatigue, and make comparisons between regorafenib dosing strategies and pre-emptive versus (vs.) reactive strategies to address PPES.

IV. Compare quality of life (QOL) between treatment arms (regorafenib dosing strategies and preemptive vs. reactive PPES strategies) as measured by the Hand and Foot Syndrome (HFS)14, Brief Fatigue Inventory (BFI), and Linear Analogue Self-Assessment (LASA) questionnaires.

TERTIARY OBJECTIVES:

I. Evaluate and compare trough minimum concentration (Cmin) pharmacokinetics (PK) during the first 2 treatment cycles for regorafenib and active metabolites M2, M5 between the low dose (dose escalation) and the standard dose cohorts, and correlate with toxicity profile.

II. Evaluate the correlation between PK parameters and tumor response/stable disease after the first two cycles.

III. Evaluate the correlation between PK parameters and PFS and OS. IV. Evaluate if trough (Cmin) concentrations are associated with patient-specific factors (such as ? but not limited to ? age and concomitant medications).

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM A1: Patients receive lower-dose regorafenib PO once daily (QD) on days 1-21 and pre-emptive clobetasol propionate given topically twice daily (BID) for 12 weeks, beginning on day 1 of regorafenib.

ARM A2: Patients receive lower-dose regorafenib PO as in Arm A1 and reactive clobetasol propionate given topically BID beginning on day 1 per physician discretion upon occurrence of PPES grade >= 1.

ARM B1: Patients receive standard dose regorafenib PO QD on days 1-21 and pre-emptive clobetasol propionate as in Arm A1.

ARM B2: Patients receive standard dose regorafenib PO as in Arm B1 and reactive clobetasol propionate as in Arm A2.

In all arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum
* Advanced or metastatic colorectal cancer with no curative options available and progression on previous standard therapy, including an EGFR inhibitor if KRAS wild-type
* Measurable or non-measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Life expectancy of >= 3 months
* Absolute neutrophil count (ANC) > 1500/mm^3 (obtained =< 7 days prior to randomization)
* Platelet count > 100,000/mm^3 (obtained =< 7 days prior to randomization)
* Hemoglobin > 9.0 g/dL (obtained =< 7 days prior to randomization)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 7 days prior to randomization)
* Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer) (obtained =< 7 days prior to randomization)
* Serum creatinine =< 1.5 x ULN (obtained =< 7 days prior to randomization)
* International normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.5 x ULN (obtained =< 7 days prior to randomization)

  * NOTE: patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists; close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care
* Alkaline phosphatase limit =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement of their cancer) (obtained =< 7 days prior to randomization)
* Negative serum pregnancy test done =< 7 days prior to randomization, for women of childbearing potential only; note: post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test; the definition of adequate contraception will be based on the judgment of the investigator
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood samples for correlative research and banking purposes

Exclusion Criteria:

* Prior treatment with regorafenib
* Major surgical procedure, open biopsy, or significant traumatic injury =< 28 days prior to randomization
* Congestive heart failure > New York Heart Association (NYHA) class 2
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months) or myocardial infarction less than 6 months prior to randomization
* Cardiac arrhythmias requiring anti-arrhythmic therapy; Note: pace makers, beta blockers, or digoxin are permitted
* Uncontrolled hypertension; (systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg despite optimal medical management)
* History of or current pheochromocytoma
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism =< 6 months prior to randomization
* Ongoing infection > grade 2 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
* Known history of chronic hepatitis B or C
* Patients with seizure disorder requiring medication
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of randomization and is clinically stable with respect to the tumor at the time of randomization; note: patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies)
* History of organ allograft (including corneal transplant)
* Evidence or history of bleeding diathesis or any hemorrhage or bleeding event > CTCAE grade 3 =< 4 weeks prior to randomization
* Non-healing wound, ulcer, or bone fracture
* Renal failure requiring hematological (hemo-) or peritoneal dialysis
* Dehydration CTCAE (version 4.0) grade >= 1
* Substance abuse, medical, psychological or social conditions that may interfere with the patient?s participation in the study or evaluation of the study results
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Persistent proteinuria of Common Toxicity Criteria (CTC) grade 3 or higher (>= 3.5 g/24 hours [hrs])
* Patients unable to swallow oral medications
* Any malabsorption condition
* Unresolved toxicity greater than CTCAE (version 4.0) grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin induced neurotoxicity =< grade 2
* Albumin levels < 2.5 g/dl
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

    * NOTE: men and women of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form (ICF) until at least 3 months after the last dose of study drug; the definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 3 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria]); note: all cancer treatments for cancers that were distinct in a primary site other than colorectal must be completed at least 3 years prior to randomization (i.e., signature date of the informed consent form)
* Pleural effusion or ascites that causes respiratory compromise (>= CTCAE version 4.0 grade 2 dyspnea)
* Concurrent anti-cancer therapy =< 4 weeks from registration (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization)
* Current use of clobetasol propionate
* Use of any herbal remedy (e.g. St. John?s wort [Hypericum perforatum])
* Patients unable to ambulate or who have amputations or paralysis of any extremity
* History of contact dermatitis to clobetasol propionate or similarly fluorinated steroids or other steroids with the propionate ester

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Bekaii-Saab, Principal Investigator — Academic and Community Cancer Research United
Locations (22):
- United States (22):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Wellmont Medical Associates Oncology and Hematology-Kingsport, Kingsport, Tennessee
  - University of Washington Medical Center, Seattle, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin

REFERENCES:
- [Derived] Bekaii-Saab TS, Ou FS, Ahn DH, Boland PM, Ciombor KK, Heying EN, Dockter TJ, Jacobs NL, Pasche BC, Cleary JM, Meyers JP, Desnoyers RJ, McCune JS, Pedersen K, Barzi A, Chiorean EG, Sloan J, Lacouture ME, Lenz HJ, Grothey A. Regorafenib dose-optimisation in patients with refractory metastatic colorectal cancer (ReDOS): a randomised, multicentre, open-label, phase 2 study. Lancet Oncol. 2019 Aug;20(8):1070-1082. doi: 10.1016/S1470-2045(19)30272-4. Epub 2019 Jun 28. PMID 31262657
- [Derived] Weinberg BA, Hartley ML, Salem ME. Precision Medicine in Metastatic Colorectal Cancer: Relevant Carcinogenic Pathways and Targets-PART 2: Approaches Beyond First-Line Therapy, and Novel Biologic Agents Under Investigation. Oncology (Williston Park). 2017 Jul 15;31(7):573-80. PMID 28712102

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy): In the regorafenib dose escalation group, the starting dose of regorafenib was 80 mg/day in week 1, 120 mg/day in week 2, and 160 mg/day in week 3 for cycle 1. Weekly incremental dose-escalation occurred if no significant drug-related toxicities (SDRTs) were observed. In cycle 2, patients received the highest tolerated dose from cycle 1. Patients also received prophylactic 0.05% clobetasol cream twice daily applied to palms and soles starting at cycle 1 day 1 for prevention of HFSR (pre-emptive strategy).
- Arm A2 (Regorafenib Dose Escalation + Reactive Strategy): In the regorafenib dose escalation group, the starting dose of regorafenib was 80 mg/day in week 1, 120 mg/day in week 2, and 160 mg/day in week 3 for cycle 1. Weekly incremental dose-escalation occurred if no significant drug-related toxicities (SDRTs) were observed. In cycle 2, patients received the highest tolerated dose from cycle 1. Patients also had the clobetasol cream applied when HFSR developed (reactive strategy).
- Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy): In the regorafenib standard dose group, the regorafenib dose schedule of 160 mg/day started on day 1 and continued for 21 every 28 days. The dose of 160 mg as the standard dose was used since it is the approved and most commonly used dose/schedule in clinical practice based on the results of randomized trials.Patients also received prophylactic 0.05% clobetasol cream twice daily applied to palms and soles starting at cycle 1 day 1 for prevention of HFSR (pre-emptive strategy).
- Arm B2 (Regorafenib Standard Dose + Reactive Strategy): In the regorafenib standard dose group, the regorafenib dose schedule of 160 mg/day started on day 1 and continued for 21 every 28 days. The dose of 160 mg as the standard dose was used since it is the approved and most commonly used dose/schedule in clinical practice based on the results of randomized trials. Patients also had the clobetasol cream applied when HFSR developed (reactive strategy).
Period: Overall Study
Arm/Group | Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy) | Arm A2 (Regorafenib Dose Escalation + Reactive Strategy) | Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy) | Arm B2 (Regorafenib Standard Dose + Reactive Strategy)
Started | 29 | 27 | 34 | 33
Completed | 28 | 26 | 33 | 29
Not Completed | 1 | 1 | 1 | 4
Not completed — Cancel | 1 | 1 | 1 | 3
Not completed — Ineligible | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The data for the pre-emptive and reactive treatment with clobatasol were pooled for the comparison of the two dosing strategies (regorafenib dose escalation group (Arms A1 + A2) versus regorafenib standard dose group (Arms B1 + B2)).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy) | Arm A2 (Regorafenib Dose Escalation + Reactive Strategy) | Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy) | Arm B2 (Regorafenib Standard Dose + Reactive Strategy) | Total
Number analyzed (Participants) | 28 | 26 | 33 | 29 | 116
Age, Continuous [Median (Full Range); unit: years] | 65 [38 to 77] | 57 [29 to 76] | 61 [32 to 78] | 62 [34 to 81] | 61 [29 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 17 | 10 | 45
  Male | 19 | 17 | 16 | 19 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 4 | 9
  White | 25 | 19 | 31 | 24 | 99
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 26 | 33 | 29 | 116
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 9 | 11 | 15 | 8 | 43
    1 | 19 | 15 | 18 | 21 | 73

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in Each Arm Who Complete 2 Cycles of Protocol Treatment and Initiate Cycle 3
Description: Fisher exact test will be used to detect a difference course 3 between arms (starting low dose [pooled arm A1 and A2] versus [vs.] standard dose [pooled arm B1 and B2]). The proportion of patients who complete 2 courses of protocol treatment and initiate course 3 will be computed by arm with its 95% confidence interval using exact method.
Time Frame: At 8 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: proportion of patients
Groups:
- Regorafenib Dose Escalation Group: In the regorafenib dose escalation group, the starting dose of regorafenib was 80 mg/day in week 1, 120 mg/day in week 2, and 160 mg/day in week 3 for cycle 1. Weekly incremental dose-escalation occurred if no significant drug-related toxicities (SDRTs) were observed. In cycle 2, patients received the highest tolerated dose from cycle 1. Patients also received prophylactic 0.05% clobetasol cream twice daily applied to palms and soles starting at cycle 1 day 1 for prevention of HFSR (pre-emptive strategy) or had the clobetasol cream applied when HFSR developed (reactive strategy).
- Regorafenib Standard Dose Group: In the regorafenib standard dose group, the regorafenib dose schedule of 160 mg/day started on day 1 and continued for 21 every 28 days. The dose of 160 mg as the standard dose was used since it is the approved and most commonly used dose/schedule in clinical practice based on the results of randomized trials.Patients also received prophylactic 0.05% clobetasol cream twice daily applied to palms and soles starting at cycle 1 day 1 for prevention of HFSR (pre-emptive strategy) or had the clobetasol cream applied when HFSR developed (reactive strategy).
Arm/Group | Regorafenib Dose Escalation Group | Regorafenib Standard Dose Group
Number analyzed (Participants) | 54 | 62
proportion of patients | 0.43 [0.29 to 0.56] | 0.26 [0.15 to 0.37]
Statistical Analysis 1: Comparison: Regorafenib Dose Escalation Group vs Regorafenib Standard Dose Group; Test type: Superiority; p = 0.0434, Fisher Exact — 1-sided; Risk Difference (RD) = 0.17, 95% CI 2-sided [0.00 to 0.34]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause and will be estimated with Kaplan-Meier survival curves and differences between regorafenib arms (A vs. B) tested using log-rank tests, though these analyses are not powered for formal non-inferiority assessments.
Time Frame: Time from randomization to death due to any cause, assessed up to 2 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib Dose Escalation Group | Regorafenib Standard Dose Group
Number analyzed (Participants) | 54 | 62
months | 9.8 [7.5 to 11.9] | 6.0 [4.9 to 10.2]
Statistical Analysis 1: Comparison: Regorafenib Dose Escalation Group vs Regorafenib Standard Dose Group; Test type: Superiority; p = 0.1241, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.47 to 1.10]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the earlier of disease progression or death due to any cause, where progressed disease (PD) is defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and will be estimated with Kaplan-Meier survival curves and differences between regorafenib arms (A vs. B) tested using log-rank tests, though these analyses are not powered for formal non-inferiority assessments.
Time Frame: Time from randomization to the earlier of disease progression or death due to any cause, where progressed disease (PD) is defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib Dose Escalation Group | Regorafenib Standard Dose Group
Number analyzed (Participants) | 54 | 62
months | 2.8 [2.0 to 5.0] | 2.0 [1.8 to 2.8]
Statistical Analysis 1: Comparison: Regorafenib Dose Escalation Group vs Regorafenib Standard Dose Group; Test type: Superiority; p = 0.3797, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.57 to 1.24]

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from randomization to disease progression, where PD is defined by RECIST 1.1 and will be estimated with Kaplan-Meier survival curves and differences between regorafenib arms (A vs. B) tested using log-rank tests, though these analyses are not powered for formal non-inferiority assessments.
Time Frame: Time from randomization to disease progression, where PD is defined by RECIST 1.1, assessed up to 2 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib Dose Escalation Group | Regorafenib Standard Dose Group
Number analyzed (Participants) | 54 | 62
months | 2.8 [1.9 to 5.7] | 2.0 [1.8 to 3.3]
Statistical Analysis 1: Comparison: Regorafenib Dose Escalation Group vs Regorafenib Standard Dose Group; Test type: Superiority; p = 0.4614, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.55 to 1.31]

5. Secondary Outcome: Cumulative (Total) Dose of Regorafenib Received by Patients in the First Two Cycles
Description: Will be summarized with descriptive statistics and compared between regorafenib arms (A vs. B).
Time Frame: Up to 8 weeks
Population: The data for the pre-emptive & reactive treatment with clobatasol were pooled for the comparison of the two dosing strategies ((Arms A1 + A2) versus (Arms B1 + B2)). There are patients off-protocol treatment during cycle 1; therefore, we do not have cycle 2 dosing information for those patients who are off-protocol treatment during cycle 1.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Regorafenib Dose Escalation Group | Regorafenib Standard Dose Group
Number analyzed (Participants) | 54 | 62
mg/day
  Cycle 1 | 91.8 (33.4) | 133.1 (34.6)
  Cycle 2: number analyzed (Participants) | 41 | 41
  Cycle 2 | 121.3 (40.0) | 117.3 (48.9)

6. Secondary Outcome: Dose Intensity of Regorafenib Received by Patients in the First Two Cycles as Measured by the Percentage of Planned Dose Received
Description: Dose intensity of regorafenib received by patients in the first two cycles as measured by the percentage (%) of planned dose received
Time Frame: Up to 8 weeks
Population: The data for the pre-emptive & reactive treatment with clobatasol were pooled for the comparison of the two dosing strategies ((Arms A1 + A2) versus (Arms B1 + B2)).
Measure: Median (Standard Deviation); unit: percentage of planned dose received
Arm/Group | Regorafenib Dose Escalation Group | Regorafenib Standard Dose Group
Number analyzed (Participants) | 54 | 62
percentage of planned dose received | 76.2 (25.3) | 76.0 (21.0)

7. Secondary Outcome: Proportion of Patients Overall and Within Each Arm Experiencing Grade 3 or 4 Hand and Foot Syndrome (HFS)
Description: Will be computed with 95% confidence intervals.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy) | Arm A2 (Regorafenib Dose Escalation + Reactive Strategy) | Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy) | Arm B2 (Regorafenib Standard Dose + Reactive Strategy)
Number analyzed (Participants) | 28 | 26 | 33 | 29
proportion of participants | 0.1786 [0.0606 to 0.3689] | 0.1154 [0.0245 to 0.3015] | 0.1515 [0.0511 to 0.3190] | 0.1724 [0.0585 to 0.3577]

8. Secondary Outcome: Quality of Life (QOL) (According to the HFS14 Total Score)
Description: Patients will be descriptively compared between treatment arms and between HFS treatment strategies (pre-emptive vs. reactive) according to self-reported outcomes given on the HFS14 questionnaire. Results from the course 1 and 2 HSF14 questionnaires will also be summarized descriptively as they relate to the pre-emptive versus reactive palmar-plantar erythrodysesthesia syndrome (PPES) strategies. Total HFS-14 score was calculated by summing the scores of all items and adjusting to 100 by applying a rule of three. Total scores have a range of 2-100, with the higher the score, the greater the QoL impairment.
Time Frame: 8 weeks
Population: Only patients that completed a post-baseline HFS14 assessment were included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy) | Arm A2 (Regorafenib Dose Escalation + Reactive Strategy) | Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy) | Arm B2 (Regorafenib Standard Dose + Reactive Strategy)
Number analyzed (Participants) | 17 | 11 | 11 | 14
score on a scale | 20.8 (19.05) | 29.5 (21.97) | 15.8 (14.65) | 21.8 (26.38)

9. Secondary Outcome: Changes in QOL (According to the Linear Analogue Self-Assessment [LASA] Questionnaire)
Description: Changes in QOL (according to the LASA questionnaire as measured by the overall QOL question) from baseline will be compared between the treatment arms using the Kruskal-Wallis test.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: LASA overall score change from baseline
Arm/Group | Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy) | Arm A2 (Regorafenib Dose Escalation + Reactive Strategy) | Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy) | Arm B2 (Regorafenib Standard Dose + Reactive Strategy)
Number analyzed (Participants) | 20 | 11 | 14 | 16
LASA overall score change from baseline | -0.9 (1.12) | -0.3 (1.42) | -0.7 (2.09) | -0.9 (1.96)
Statistical Analysis 1: Comparison: Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy) vs Arm A2 (Regorafenib Dose Escalation + Reactive Strategy) vs Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy) vs Arm B2 (Regorafenib Standard Dose + Reactive Strategy); Test type: Superiority; p = 0.7319, Kruskal-Wallis

10. Other Pre Specified Outcome: Pharmacokinetics (PK) Parameters of Regorafenib Using Liquid Chromatography Mass Spectrometry
Description: After quantitation, the average trough concentration, calculated from all available data, will be calculated. This average trough concentration will be correlated with toxicity and efficacy endpoints. Further descriptive characteristics of the pharmacokinetics will also be calculated, an example includes (but is not limited to) within-patient variability in the trough concentrations pharmacokinetic parameters will also be calculated, both overall and within courses, as a ratio of the maximum:minimum value.
Time Frame: Baseline, prior to treatment, days 7, 14, and 21 prior to treatment (course 1), and days 1 and 21 prior to treatment (course 2)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during the active monitoring phase (weekly during Cycles 1 and 2, then every 4 weeks until progression); up to 2 years. The total study duration (accrual and follow-up) is expected to be approximately 2 years.
Description: Each CTCAE term is a representation of a specific event used for medical documentation & analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for non-cancel patients. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Groups:
- Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy): In the regorafenib standard dose group, the regorafenib dose schedule of 160 mg/day started on day 1 and continued for 21 every 28 days. The dose of 160 mg as the standard dose was used since it is the approved and most commonly used dose/schedule in clinical practice based on the results of randomized trials. Patients also received prophylactic 0.05% clobetasol cream twice daily applied to palms and soles starting at cycle 1 day 1 for prevention of HFSR (pre-emptive strategy).
Arm/Group | Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy) | Arm A2 (Regorafenib Dose Escalation + Reactive Strategy) | Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy) | Arm B2 (Regorafenib Standard Dose + Reactive Strategy)
All-Cause Mortality (participants affected / at risk) | 0/28 | 3/26 | 3/33 | 2/30
Serious Adverse Events (participants affected / at risk) | 4/28 | 10/26 | 10/33 | 10/30
Other Adverse Events (participants affected / at risk) | 28/28 | 24/26 | 31/33 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy) (N=28) | Arm A2 (Regorafenib Dose Escalation + Reactive Strategy) (N=26) | Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy) (N=33) | Arm B2 (Regorafenib Standard Dose + Reactive Strategy) (N=30)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A1 (Regorafenib Dose Escalation + Pre-emptive Strategy) (N=28) | Arm A2 (Regorafenib Dose Escalation + Reactive Strategy) (N=26) | Arm B1 (Regorafenib Standard Dose + Pre-emptive Strategy) (N=33) | Arm B2 (Regorafenib Standard Dose + Reactive Strategy) (N=30)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 8 (15) | 7 (10) | 6 (8)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 3 (3) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 14 (30) | 10 (20) | 17 (37) | 10 (24)
Dry mouth (Gastrointestinal disorders) | 2 (7) | 1 (1) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 4 (5) | 5 (7) | 5 (7)
Nausea (Gastrointestinal disorders) | 8 (16) | 12 (21) | 16 (43) | 13 (17)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (5)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (7) | 7 (8) | 9 (12) | 5 (6)
Chills (General disorders) | 1 (2) | 1 (3) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 25 (72) | 20 (53) | 26 (83) | 27 (72)
Fever (General disorders) | 1 (2) | 0 (0) | 1 (1) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (4)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 4 (4) | 6 (13) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (4) | 4 (4) | 7 (13) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 5 (8) | 8 (16) | 8 (9)
Blood bilirubin increased (Investigations) | 3 (5) | 5 (5) | 9 (10) | 9 (10)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 3 (4)
Investigations - Other, specify (Investigations) | 1 (8) | 1 (1) | 2 (5) | 3 (4)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (5) | 2 (3) | 4 (6)
Platelet count decreased (Investigations) | 4 (4) | 2 (3) | 6 (8) | 2 (2)
Weight loss (Investigations) | 2 (3) | 3 (9) | 6 (9) | 5 (5)
White blood cell decreased (Investigations) | 1 (2) | 1 (1) | 3 (3) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (11) | 6 (7) | 6 (10) | 13 (20)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6) | 2 (2) | 3 (5) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3) | 0 (0) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 3 (4) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (8) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 1 (2) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (5) | 3 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (4) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (6) | 3 (7) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6) | 1 (1) | 4 (8) | 2 (4)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (7) | 5 (5) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (11) | 4 (8) | 5 (6) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (9) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1) | 2 (7) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 18 (37) | 17 (43) | 22 (61) | 22 (42)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (16) | 2 (3) | 8 (12) | 8 (11)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 21 (46) | 14 (36) | 17 (62) | 19 (44)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT02368886/Prot_SAP_000.pdf